CLINICAL TRIAL: NCT04967105
Title: Intraoperative Renal Desaturation and Postoperative Acute Kidney Injury in Elderly Patients Undergoing Liver Resection: a Prospective Cohort Study
Brief Title: Intraoperative Renal Desaturation and Postoperative Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-003
Record Dates: First submitted 2021-07-12; First posted 2021-07-19 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Acute Kidney Injury
Keywords: liver resection; elderly; renal oxygen saturation; near-infrared spectroscopy
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients following liver resection: elderly patients (aged ≥60 years) scheduled for any type of liver resection due to benign or malignant hepatobiliary diseases
  Interventions: Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Near-infrared spectroscopy — Before the induction of anesthesia, NIRS sensors were placed on both sides of the flank area that overlies the kidney to monitor renal SO2, whose alteration trends over time during operation will be recorded and evaluated in later analysis.

SUMMARY:
The aim of this study is to investigate the changes in renal regional oxygen saturation (rSO2) monitored by near-infrared spectroscopy (NIRS) and its relationship with the occurrence of postoperative AKI.

DETAILED DESCRIPTION:
Postoperative acute kidney injury (AKI) is a severe complication after liver resection and contributes to increased morbidity and mortality.

Advanced age reduces renal autoregulatory capacity due to physiological and functional changes, thus render the elderly to suffer postoperative AKI and probably the consequent chronic kidney disease. Thus, it is essential to identify those patients at high risk to develop postoperative AKI to optimize perioperative prevention and protection strategies.

Despite the multiple risk factors and potential mechanisms that have been identified, the diagnosis of postoperative AKI depending on serum creatinine changes have been delayed for early identification of postoperative AKI. It is of great interest to develop target strategies for close motoring of renal function.

This study is a prospective cohort study to investigate the associations between intraoperative renal desaturation measured by NIRS and postoperative AKI. The investigators intend to access the optimal threshold values of renal rSO2 for predicting postoperative AKI. Desaturation of renal rSO2 will be defined by the severity and duration of NIRS values during the surgical process. The principal clinical outcome of the study is postoperative AKI, defined as an absolute increase in serum creatinine of 0.3 mg/dL within 48 hours or a 1.5-fold increase from preoperative baseline within seven days after surgery, according to the Kidney Disease: Improving Global Outcomes (KDIGO) criterion.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (defined as 60 years of age or older) scheduled for elective liver resection

Exclusion Criteria:

* Emergency surgery
* Liver transplantation
* Preoperative hemodialysis
* BMI > 30
* Renal depth (distance from the capsule of the kidney to the skin surface) > 4 cm
* Unable or failed to sign the informed consent

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 60 years who intend to receive elective hepatectomy surgeries
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Postoperative 7 days
  Postoperative acute kidney injury is defined according to the KDIGO criterion

SECONDARY OUTCOMES:
Death before and 30 days after discharge | 30 days after discharge
  Collection of clinical data in the medical record and follow-up update through telephone
Length of hospital stay | Postoperative 30 days
  Collection of clinical data in the medical record

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided